CLINICAL TRIAL: NCT06572826
Title: A framEwork for aN InteGrated assessMent of cArdiac Rehabilitation Programs in Patients Acutely Managed for Cardiogenic Shock - ENIGMA-shock
Brief Title: Cardiac Rehabilitation in Patients Acutely Managed for Cardiogenic Shock (ENIGMA)
Acronym: ENIGMA
Status: Recruiting | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Ospedale Civile Ss. Antonio e Biagio e Cesare Arrigo, Alessandria, Italy (Unknown); Azienda Ospedaliera Brotzu (Other); Azienda Ospedaliera OO.RR. S. Giovanni di Dio e Ruggi D'Aragona (Other); ASST Grande Ospedale Metropolitano Niguarda, Milano, Italy (Unknown)
Responsible Party: Sponsor
Other Study IDs: ENIGMA
Record Dates: First submitted 2024-08-21; First posted 2024-08-27 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Cardiogenic Shock
Keywords: Cardiogenic Shock; Rehabilitation
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiogenic Shock: Study population: All consecutive patients with a clinical diagnosis of Cardiogenic Shock enrolled in the Altshock registry will be included.
  Interventions: Other: Cardiac Rehabilitation intervention

INTERVENTIONS:
Other: Cardiac Rehabilitation intervention — The cardiac rehabilitation program for post-CS patients includes respiratory physiotherapy, muscle strengthening and endurance training such as walking, treadmill exercises, and cycling, all tailored to the patient's capabilities. Cardiovascular training involves interval and continuous aerobic exercises to improve heart function. The program emphasizes secondary prevention strategies, including lifestyle changes and medication management. Neuromotor rehabilitation addresses sarcopenia and polyneuropathies through targeted exercises like balance training, gait retraining, and the use of advanced technologies like functional electrical stimulation (FES), robotic devices, and virtual/augmented reality. Cognitive-behavioral therapy (CBT) helps manage the psychological effects of severe cardiovascular events. The program also includes speech and occupational therapy, planning for home reintegration, and telerehabilitation to ensure long-term recovery.

SUMMARY:
This is a prospective and retrospective multicentre study conducted under the scientific coordination of the IRCCS Fondazione Don Gnocchi and funded by the Italian Ministry of Health (PNRR-MCNT2-2023-12377767). Using the Altshock registry, the largest multicentre Cardiogenic Shock (CS) registry in Italy, which currently has registered more than 1,000 CS patients across Italy, we will recruit patients to: (1) provide a granular assessment of post-acute phase programmes, patients' functional disability, return to work and quality of life, including specific reference to gender; (2) implement specific pathways of care in the post-acute phase; (3) provide a multidimensional assessment, thus validating an innovative model in comparison with the traditional pathway, defining the potential benefits to and impact on economic efficiency and the general sustainability of this therapeutic trajectory.

DETAILED DESCRIPTION:
Study Population: The study will include all consecutive Cardiogenic Shock (CS) patients from the Altshock registry. The primary outcome is all-cause death and readmission-free survival at 6 months and 1 year post-ICU discharge. Secondary outcomes include functional recovery measured by illness severity (using the Medical Research Council Scale and electromyography if needed), disease-specific PROM (Kansas City Cardiomyopathy Questionnaire), and a chronic condition PROM (Long-Term Conditions Questionnaire) at 6 months.

Sample Size: An estimated cohort of 2000 CS patients, with around 1240 survivors, will be studied. This sample allows us to detect a 10% difference in death and readmission-free survival rates between those receiving post-acute care services and those who do not, with 80% power and a 5% significance level.

Validation and Assessment: A mixed-method approach will validate the innovative care model, incorporating clinical data, health economics, and professional perceptions. Key performance indicators and a RACI matrix will guide the implementation, with a focus on short- and long-term organizational impacts, economic benefits, and healthcare professional perceptions.

Data Analysis: Quantitative variables will be analyzed using standard statistical methods, and survival analysis will compare groups using Kaplan-Meier curves and log-rank tests. Multivariable Cox models will assess the impact of post-acute care services on outcomes. Economic analyses will involve cost-effectiveness and budget impact assessments.

Rehabilitation Intervention: Post-acute care, including cardiac and neuromotor rehabilitation, is critical for CS patients to prevent complications and rehospitalization. The rehabilitation program will include respiratory physiotherapy, muscle strengthening, endurance training, cardiovascular exercises, and secondary prevention strategies. Neuromotor rehabilitation will address sarcopenia and polyneuropathies with targeted exercises and advanced technologies like robotics and FES.

Expected Outcomes: The ENIGMA project aims to improve CS patient outcomes by transforming post-acute care, reducing mortality, enhancing quality of life, and proving the cost-effectiveness and sustainability of innovative care pathways.

ELIGIBILITY:
Inclusion Criteria:

• All consecutive patients with a clinical diagnosis of Cardiogenic Shock.

Exclusion Criteria:

• Refusal to give informed consent.

Ages: 18 Years to 110 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All consecutive patients with Cardiogenic Shock (CS) will be included. The deferred consent is admitted for non-competent patients.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-08-31 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
All-cause of death | 1 Year
  Incidence of all-cause death
Readmission in hospital for any cause | 1 Year
  Incidence of readmission

SECONDARY OUTCOMES:
Severity of critical illness polyneuropathy | 6-months
  Assessment using clinical evaluation (using the Medical Research Council Scale for Muscle Strength), with electromyography and nerve conduction if required
Disease-specific PROM | 6-Months
  The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a specialized tool designed to assess the health-related quality of life in patients with heart failure. It measures the physical, social, and emotional impacts of heart failure, providing insights into the effectiveness of treatments and guiding clinical decisions.
Chronic-condition PROM | 6-months
  standardized by the Food and Drug Administration and the Oxford Patient-Reported Outcomes Group's Long-Term Conditions Questionnaire
PREMS: patient's opinion regarding their clinical service. | 6-months
  Patients will be questioned about the clinical service received. The items explored will be coordination and integration of care; information, communication, and education; physical comfort; emotional support; welcoming and involvement of family and friends; transition and continuity; and access to care. Patients will define every item in terms of low quality, moderate quality and high quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Don Gnocchi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Rab T, Ratanapo S, Kern KB, Basir MB, McDaniel M, Meraj P, King SB 3rd, O'Neill W. Cardiac Shock Care Centers: JACC Review Topic of the Week. J Am Coll Cardiol. 2018 Oct 16;72(16):1972-1980. doi: 10.1016/j.jacc.2018.07.074. PMID 30309475
- [Result] Luscher TF, Thiele H. Cardiogenic shock: do we need a paradigm shift? Eur Heart J. 2024 Oct 14;45(39):4178-4180. doi: 10.1093/eurheartj/ehae425. No abstract available. PMID 38985011
- [Result] van Diepen S, Katz JN, Albert NM, Henry TD, Jacobs AK, Kapur NK, Kilic A, Menon V, Ohman EM, Sweitzer NK, Thiele H, Washam JB, Cohen MG; American Heart Association Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; Council on Quality of Care and Outcomes Research; and Mission: Lifeline. Contemporary Management of Cardiogenic Shock: A Scientific Statement From the American Heart Association. Circulation. 2017 Oct 17;136(16):e232-e268. doi: 10.1161/CIR.0000000000000525. Epub 2017 Sep 18. PMID 28923988
- [Result] Kapur NK, Kanwar M, Sinha SS, Thayer KL, Garan AR, Hernandez-Montfort J, Zhang Y, Li B, Baca P, Dieng F, Harwani NM, Abraham J, Hickey G, Nathan S, Wencker D, Hall S, Schwartzman A, Khalife W, Li S, Mahr C, Kim JH, Vorovich E, Whitehead EH, Blumer V, Burkhoff D. Criteria for Defining Stages of Cardiogenic Shock Severity. J Am Coll Cardiol. 2022 Jul 19;80(3):185-198. doi: 10.1016/j.jacc.2022.04.049. PMID 35835491
- [Result] Mueller S, Winzer EB, Duvinage A, Gevaert AB, Edelmann F, Haller B, Pieske-Kraigher E, Beckers P, Bobenko A, Hommel J, Van de Heyning CM, Esefeld K, von Korn P, Christle JW, Haykowsky MJ, Linke A, Wisloff U, Adams V, Pieske B, van Craenenbroeck EM, Halle M; OptimEx-Clin Study Group. Effect of High-Intensity Interval Training, Moderate Continuous Training, or Guideline-Based Physical Activity Advice on Peak Oxygen Consumption in Patients With Heart Failure With Preserved Ejection Fraction: A Randomized Clinical Trial. JAMA. 2021 Feb 9;325(6):542-551. doi: 10.1001/jama.2020.26812. PMID 33560320
- [Result] Molloy C, Long L, Mordi IR, Bridges C, Sagar VA, Davies EJ, Coats AJ, Dalal H, Rees K, Singh SJ, Taylor RS. Exercise-based cardiac rehabilitation for adults with heart failure. Cochrane Database Syst Rev. 2024 Mar 7;3(3):CD003331. doi: 10.1002/14651858.CD003331.pub6. PMID 38451843
- [Result] Anderson L, Oldridge N, Thompson DR, Zwisler AD, Rees K, Martin N, Taylor RS. Exercise-Based Cardiac Rehabilitation for Coronary Heart Disease: Cochrane Systematic Review and Meta-Analysis. J Am Coll Cardiol. 2016 Jan 5;67(1):1-12. doi: 10.1016/j.jacc.2015.10.044. PMID 26764059
- [Result] Balady GJ, Ades PA, Bittner VA, Franklin BA, Gordon NF, Thomas RJ, Tomaselli GF, Yancy CW; American Heart Association Science Advisory and Coordinating Committee. Referral, enrollment, and delivery of cardiac rehabilitation/secondary prevention programs at clinical centers and beyond: a presidential advisory from the American Heart Association. Circulation. 2011 Dec 20;124(25):2951-60. doi: 10.1161/CIR.0b013e31823b21e2. Epub 2011 Nov 14. No abstract available. PMID 22082676
- [Result] Yang T, Li Z, Jiang L, Wang Y, Xi X. Risk factors for intensive care unit-acquired weakness: A systematic review and meta-analysis. Acta Neurol Scand. 2018 Aug;138(2):104-114. doi: 10.1111/ane.12964. Epub 2018 May 29. PMID 29845614
- [Result] Lavie CJ, Ozemek C, Carbone S, Katzmarzyk PT, Blair SN. Sedentary Behavior, Exercise, and Cardiovascular Health. Circ Res. 2019 Mar;124(5):799-815. doi: 10.1161/CIRCRESAHA.118.312669. PMID 30817262
- [Result] Aburub A, Darabseh MZ, Badran R, Shurrab AM, Amro A, Degens H. The Application of Robotics in Cardiac Rehabilitation: A Systematic Review. Medicina (Kaunas). 2024 Jul 18;60(7):1161. doi: 10.3390/medicina60071161. PMID 39064590
- [Derived] Morici N, Foglia E, Ferrario L, Pedersini P, Corda M, Ravera A, Oreni LM, Cusmano I, Garatti L, Toccafondi A, Sacco A, Oliva F, Garascia A, Frea S, Pistono M, Aschieri D, Tavazzi G, Pappalardo F. ENIGMA-shock: protocol for a study framEwork for aN InteGrated assessMent of cArdiac rehabilitation programmes in patients acutely managed for cardiogenic shock. BMJ Open. 2025 Feb 12;15(2):e092790. doi: 10.1136/bmjopen-2024-092790. PMID 39938955